CLINICAL TRIAL: NCT06704984
Title: The Effectiveness of WeChat Public Account Intervention Based on the IMB Model Among College Students With Internet Addiction: A Randomized Controlled Trial
Brief Title: Effectiveness of WeChat Public Account Intervention Based on the IMB Model for College Students With Internet Addiction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shihaiyan Shi (Other)
Responsible Party: Sponsor-Investigator, Shihaiyan Shi, Principal Investigator, Anhui Medical University
Organization: Anhui Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20190495
Record Dates: First submitted 2024-11-09; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Internet Addiction
Keywords: IMB model; Internet addiction; WeChat public accounts; Randomized controlled trial; Intervention
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Intervention Model Description: Intervention Group: Intervention based on the IMB model through WeChat official account
  Control Group: No intervention, maintaining normal life and study status
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention group: A six-week intervention leveraging an online WeChat public account was implemented, integrating the IMB (Information-Motivation-Behavioral Skills) model into its design. Drawing from literature analysis, the intervention plan was structured into three distinct modules: information, motivation, and behavioral skills. The comprehensive intervention encompassed disseminating knowledge on Internet addiction, identifying and avoiding triggers, fostering withdrawal motivation, imparting coping strategies for cravings and challenging situations, enhancing self-efficacy, and facilitating access to personal and social support. Participants who followed the WeChat public account received automated push notifications containing articles or videos every two days. Throughout the intervention period, engagement was monitored by tracking the readership of the sent content through the WeChat public account's backend data.
  Interventions: Behavioral: Intervention Name: WeChat Intervention Based on the IMB Model
- Control group (No Intervention): Control group: without any intervention, maintain normal life and study state.

INTERVENTIONS:
Behavioral: Intervention Name: WeChat Intervention Based on the IMB Model — A six-week intervention leveraging an online WeChat public account was implemented, integrating the IMB (Information-Motivation-Behavioral Skills) model into its design. Drawing from literature analysis, the intervention plan was structured into three distinct modules: information, motivation, and behavioral skills. The comprehensive intervention encompassed disseminating knowledge on Internet addiction, identifying and avoiding triggers, fostering withdrawal motivation, imparting coping strategies for cravings and challenging situations, enhancing self-efficacy, and facilitating access to personal and social support. Participants who followed the WeChat public account received automated push notifications containing articles or videos every two days. Throughout the intervention period, engagement was monitored by tracking the readership of the sent content through the WeChat public account's backend data.
  Arms: Intervention group

SUMMARY:
Objective:

The investigators want to see if a WeChat program can help college students use the internet less and feel better.

Methods:

The investigators picked 226 students who use the internet too much. The investigators put 113 in a group that used a special WeChat program for six weeks. The other 113 did nothing different. The investigators checked how much they used the internet, slept, and how they felt before and after.

Interventions:

The WeChat program gave students info, motivation, and skills to cut down on internet use. It sent them articles and videos every two days.

Data Collection and Outcome Measures:

The investigators used a test to see how much students were addicted to the internet. The investigators also looked at their internet time, sleep, and feelings. The investigators used math tricks to see if the program worked.

Brief Summary:

This study checks if a WeChat program can help students with internet addiction. It teaches them about their habits and how to change them.

DETAILED DESCRIPTION:
Background:

With the rise of digital technology, internet addiction has become a significant concern among college students, affecting their academic performance and mental health. The Information-Motivation-Behavioral Skills (IMB) model has shown promise in understanding and addressing health behaviors, including addiction.

Objective:

The primary objective of this study is to evaluate the effectiveness of a WeChat public account intervention based on the IMB model in reducing internet addiction among college students. The study also aims to explore the underlying mechanisms that lead to changes in addictive behaviors, contributing to the development of a new online treatment model for internet addiction.

Methods:

A total of 226 college students diagnosed with internet addiction were recruited and randomly assigned to either an intervention group (n=113) or a control group (n=113) using stratified randomization based on gender. The intervention group participated in a structured six-week program that leveraged a WeChat public account to deliver content designed to educate about internet addiction, identify triggers, enhance motivation to change, and improve behavioral skills. The control group maintained their regular routines without any intervention. Data were collected before and after the intervention period using standardized measures, including the Internet Addiction Test (IAT), and assessed for internet usage time, sleep duration, sleep quality, and somatic-psychological symptoms.

Interventions:

The intervention was structured around three modules: information, motivation, and behavioral skills. Participants in the intervention group received automated push notifications with articles or videos every two days through the WeChat public account. The content was designed to provide knowledge about internet addiction, strategies to cope with cravings, and methods to enhance self-efficacy and access to support. The intervention was monitored through the account's backend data to track engagement.

Data Collection and Outcome Measures:

The main outcome measure was the IAT scale score, which assesses the severity of internet addiction. Secondary outcomes included changes in internet usage time, sleep duration, sleep quality, and somatic-psychological symptoms. Data were analyzed using Generalized Linear Mixed Models (GLMM) and Generalized Estimating Equations (GEE) to evaluate the impact of the intervention and to identify differences pre- and post-intervention.

Significance:

The findings of this study could provide valuable insights into the effectiveness of digital interventions for internet addiction and contribute to the development of targeted prevention and treatment strategies for college students.

ELIGIBILITY:
Inclusion Criteria:

* College students diagnosed with Internet addiction, as evidenced by an IAT scale score of 40 or above.
* Age range between 18 and 24 years.
* Use WeChat software.
* Good physical health, capable of completing the whole process of the study.
* Voluntary participation with a signed Informed Consent form.

Exclusion Criteria:

* Presence of any mental illness or cognitive impairment.
* Current or impending receipt of psychological or pharmacological treatment for a mental health condition.
* Circumstances that would hinder participation, such as internships, suspensions, or other reasons for absence from school.
* Refusal to participate in the study.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 226 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2023-06-19 (Actual)

PRIMARY OUTCOMES:
Internet Addiction | From enrollment to the end of treatment at 6 weeks
  Internet Addiction Measurement Tool: 20-item Internet Addiction Test (IAT) Description: Scores range from 20 to 100, with higher scores indicating a more severe level of internet addiction (20-39: no addiction, 40-69: mild addiction, ≥70: moderate to severe addiction).

SECONDARY OUTCOMES:
Internet Usage Time | From enrollment to the end of treatment at 6 weeks
  Internet Time Measurement: Minutes Description: Higher values indicate longer internet usage time.
Sleep Duration | From enrollment to the end of treatment at 6 weeks.
  Sleep Duration Measurement: Minutes Description: Higher values indicate longer sleep time
Sleep Quality | From enrollment to the end of treatment at 6 weeks.
  Sleep Quality Measurement Tool: Pittsburgh Sleep Quality Index (PSQI) Description: Scores range from 0 to 3, with higher scores indicating poorer sleep quality. This RCT includes only the components of sleep quality and sleep duration.
Somatic-Psychological Symptoms | From enrollment to the end of treatment at 6 weeks.
  Somatic-Psychological Symptoms Measurement Tool: Symptom Checklist Description: Binary outcomes indicating the presence or absence of specific symptoms, including Dizziness, Eye Discomfort, Gastrointestinal Problems, Low Mood, and Anxiety.

OTHER OUTCOMES:
Knowledge of Internet Addiction (Information) | From enrollment to the end of treatment at 6 weeks.
  Knowledge of Internet Addiction (Information) Measurement Tool: Self-designed questionnaire based on "Knowledge and Attitude of Internet Addiction" by Huang Yurong et al.
  Description: Comprises 10 judgment questions with a scoring system (1 point for correct, 0 for incorrect/unclear), including reverse scoring for items 3, 4, 7, and 9 to minimize bias. Total score ranges from 0 to 10, with higher scores indicating better knowledge.
Motivation for Internet Addiction Improvement (Motivation) | From enrollment to the end of treatment at 6 weeks.
  Motivation for Internet Addiction Improvement (Motivation):
  Measurement Tool: Treatment Self-Regulation Questionnaire (TSRQ), Chinese version by Zhou Chenxi et al.
  Description: 15-item questionnaire with a 7-point Likert scale, scoring from 15 to 105. Higher scores indicate stronger motivation for treatment.
Internet Control Self-Efficacy (Behavioral Skills) | From enrollment to the end of treatment at 6 weeks.
  Internet Control Self-Efficacy (Behavioral Skills) Measurement Tool: Internet Control Self-Efficacy Questionnaire (ICSQ) by Luo et al.
  Description: 12-item questionnaire focusing on time management, task control, and purpose clarity. 4-point Likert scale, total score from 12 to 48. Higher scores indicate greater self-efficacy in controlling internet use.

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bai Y, Qu J, Li D, Yin H. Neural basis underlying the relation between internet addiction tendency and sleep quality: The intrinsic default-mode network connectivity pathways. Int J Psychophysiol. 2024 Jan;195:112264. doi: 10.1016/j.ijpsycho.2023.112264. Epub 2023 Nov 15. PMID 37977269
- [Background] Aziz M, Chemnad K, Al-Harahsheh S, Abdelmoneium AO, Bagdady A, Hassan DA, Ali R. The influence of adolescents essential and non-essential use of technology and Internet addiction on their physical and mental fatigues. Sci Rep. 2024 Jan 19;14(1):1745. doi: 10.1038/s41598-024-51655-x. PMID 38242916